CLINICAL TRIAL: NCT01134016
Title: Determine MTD and to Evaluate PK, Safety/Tolerability and Efficacy Profiles of Antroquinonol (Hocena®) in NSCLC Patients Refractory to Conventional Treatment Modalities
Brief Title: Determine MTD and to Evaluate pk, Safety/Tolerability and Efficacy Profiles of Hocena® in NSCLC Subjects
Acronym: Hocena
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Collaborators: PharmaNet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOLANTA20090911
Record Dates: First submitted 2010-05-14; First posted 2010-05-31 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2014-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — antroquinonol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antroquinonol (Experimental): 6 dose levels, Dose Level 1 (4 weeks) : 50 mg Antroquinonol; Dose Level 2 (4 weeks) : 100mg Antroquinonol; Dose Level 3 (4 weeks) : 200mg Antroquinonol; Dose Level 4 (4 weeks) : 300mg Antroquinonol; Dose Level 5 (4 weeks) : 450mg Antroquinonol; Dose Level 6 (4 weeks) : 600mg Antroquinonol.
  A maximum of 36 patients were planned based on a criteria of a maximum of 6 patients per cohort: 1 to 6 patients were planned for each dose group in the accelerated phase; 3 to 6 patients for each dose group in the standard phase .
  The method of dose escalation in the accelerated titration phase continued to the next higher dose level until a patient experienced MT or a DLT. Standard titration phase start with 3+3 patients. Dose escalation proceeded sequentially between cohorts.
  Interventions: Drug: Antroquinonol

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol was taken orally, daily, within 15 minutes after a breakfast at the assigned dose level: 50, 100, 200, 300, 450, 600 mg/day for 4 weeks.
  Dose Level 1 (4 weeks) : 50 mg Antroquinonol; Dose Level 2 (4 weeks) : 100mg Antroquinonol; Dose Level 3 (4 weeks) : 200mg Antroquinonol; Dose Level 4 (4 weeks) : 300mg Antroquinonol; Dose Level 5 (4 weeks) : 450mg Antroquinonol; Dose Level 6 (4 weeks) : 600mg Antroquinonol.
  The accelerated phase ended when either 1 DLT or MT was observed to start standard phase. Study ended when reach the highest dose level or DLT founded.
  Other Names: Hocena

SUMMARY:
A phase I study to determine the maximum tolerable dose (MTD) and to evaluate pharmacokinetic, safety/tolerability and efficacy profiles of antroquinonol (Hocena®) in non-small cell lung cancer (NSCLC) subjects refractory to conventional treatment modalities

DETAILED DESCRIPTION:
1. Antroquinonol, a novel cyclohexenone compound, is a purified compound from extract of Antrodia camphorata.
2. The pharmacological effects of antroquinonol were postulated to exert its antitumorigenesis effects through interactions to primary targets of epidermal growth factor receptor (EGFR)/Akt/mitogen-activated protein kinase (MAPK).
3. In vivo study in NOD/SCID mice with A549 subcutaneous xenografts consistently showed tumor growth suppression after 2 weeks of oral 30 and 60 mg/kg antroquinonol treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years.
2. Diagnosed stage III/IV NSCLC. The grading is determined according to the Tumor-Node-Metastasis (TNM) staging system for lung cancer.
3. Patients with histologically or cytologically proven primary NSCLC with adenocarcinoma or mixed cell type with adenocarcinoma, who have failed on standard treatments.
4. With progressive tumor after two lines of chemotherapy (including one platinum-based) and 1 EGFR-targeted therapy if patient is identified with EGFR mutation or his/her EGFR mutation status is unknown OR having refused further currently approved treatment modalities.
5. Life expectancy ≥ 3 months.
6. Within 1 week of planned first study treatment day, adequate hematopoietic functions are presented: Total white blood cell (WBC) ≥ 3500 cells/mm3 Hemoglobin (Hb) ≥ 9.0 g/dL Platelets ≥ 100,000 cells/mm3 Absolute neutrophil count (ANC) ≥ 1500 /mm3
7. Within 1 week of planned first study treatment day, adequate hepatic and renal functions are presented: Total bilirubin ≤2.0 mg/dLGOLANTA20090911, Amendment 4/v. 1.0/ 13 October 2010 AST ≤ 3 × upper limit of normal (ULN); patients with liver metastasis: AST ≤ 5 × ULN ALT ≤ 3 × ULN; patients with liver metastasis: ALT ≤ 5 × ULN Creatinine ≤ 1.5 mg/dL
8. Must have recovered from toxicities of previous anti-cancer treatments to grade 1 NCI-CTC or better, except for alopecia.
9. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2.
10. Female patient with childbearing potential confirmed of not being pregnant at the screening; and informed that effective contraception must be used during the entire treatment period of this study and for 6 months after exiting from the study.
11. Given signed and dated written informed consent form.

Exclusion Criteria:

1. Primary major surgery < 4 weeks prior to the planned first study treatment day.
2. Lactating, pregnant or plans to be become pregnant.
3. Except for alopecia, recovered from any previous treatments to a grade 1 or less prior to the planned first study treatment day.
4. With active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal ulcers, or medical conditions that may significantly affect adequate absorption of investigational product.
5. Within 5 years, prior history of malignancy other than NSCLC, except cervical carcinoma in situ and basal or squamous cell skin carcinoma.
6. Known allergic to antroquinonol or its formulation excipients.
7. Within 14 days of planned first study treatment day, exposed to any drug(s) known to be significant CYP2C19, 3A4, 2C8, and 2E1, inhibitor or activator.
8. With conditions judged by the investigator as unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Woei-Yau Kao, M.D., Principal Investigator — Tri-Service General Hospital; Yu-Chin Lee, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (2):
- Taiwan (2):
  - Tri-Service General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participlant data(IPD).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 patients were enrolled and treated: 1 patient each received 50, 100, 200, and 300 mg, 4 patients received 450 mg, and 5 patients received 600 mg. The recruitment period is from 19 Jan 2010 to 13 Dec 2012 in list two medical center, Taiwan.
Pre-assignment Details: This was an open-label, non-randomized, dose escalation, PK study to determine the MTD and DLTs and to explore the PK, safety/tolerability, and preliminary efficacy profiles of antroquinonol.
Groups:
- Antroquinonol: Safety dose finding from 50mg to 600mg
  Antroquinonol : Dosage form: 50 mg and 100 mg capsules
  Dosage levels: 50 mg, 100 mg, 200 mg, 300mg, 450mg and 600mg ( 6 cohorts)
  Frequency: take daily for 4 weeks per subject per dosage level
Period: Overall Study
Arm/Group | Antroquinonol
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: A total of 13 patients were enrolled in this study
Arm/Group | Antroquinonol
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 13
Height [Mean (Full Range); unit: cm] | 159.76 [143 to 172]
Weight [Mean (Full Range); unit: Kg] | 64.57 [45.7 to 79.2]
BMI [Mean (Full Range); unit: kg/m^2] | 25.214 [21.15 to 32.97]

OUTCOME MEASURES:

1. Primary Outcome: To Determind the Maximum Tolerable Dose for Antroquinonol
Description: The study design consisted of 2 phases, the accelerated titration phase and the standard titration phase.
  During the accelerated titration phase, patients were enrolled in a cohort of 1 new patient for each dose level and treated for 4 weeks at that level. Any DLT or instance of MT during any 4 week treatment at any dose level led to the initiation of standard titration (3+3) phase.
  If none of the first 3 patients experienced any DLT, then dose escalation proceeded for the next cohort of patients. If 1 of 3 patients developed DLT, the cohort was expanded to at most 6 patients (another 3 patients added subsequently). If exactly 1 of the 6 patients experienced DLT, then escalation to the next dose level occurred. If more than 1 patient developed DLT in any dose cohort, the dose escalation was withheld and the prior dose level was considered as the MTD unless the present dose level was level 1
Time Frame: DLT is to be observed during 4 week period
Population: Intent-to-Treat (ITT) Population: All patients who received at least 1 dose of antroquinonol.
Measure: Number; unit: mg
Groups:
- Antroquinonol: Maximum Tolerable Dose for Antroquinonol
Arm/Group | Antroquinonol
Number analyzed (Participants) | 13
mg | 600

2. Secondary Outcome: Tmax After Dose
Description: Pharmacokinetic samples will be obtained from all the patients in each dose cohort treated in all phases of the study. Patients will only be sampled during their first treatment cycle only. Individual serum concentration versus (vs) time curves were plotted in 1 graph by dose level on both linear/linear and log10/linear scales. Mean serum concentration vs time curves were also presented in 1 graph for dose levels on both linear/linear and log10/linear scales.
Time Frame: 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 1&28
Measure: Median (Full Range); unit: hours
Groups:
- Tmax Day1: 50mg; Tmax Day 1: 100 mg; Tmax Day 1: 200mg; Tmax Day 1: 300mg; Tmax Day 1: 450mg; Tmax Day 1 :600 mg; Tmax Day 28: 50mg; Tmax Day 28: 100mg; Tmax Day 28: 200 mg; Tmax Day 28: 300mg; Tmax Day 28: 450mg; Tmax Day 28: 600mg: Patient represent the time to reach the maximum plasma concentration after dose
Arm/Group | Tmax Day1: 50mg | Tmax Day 1: 100 mg | Tmax Day 1: 200mg | Tmax Day 1: 300mg | Tmax Day 1: 450mg | Tmax Day 1 :600 mg | Tmax Day 28: 50mg | Tmax Day 28: 100mg | Tmax Day 28: 200 mg | Tmax Day 28: 300mg | Tmax Day 28: 450mg | Tmax Day 28: 600mg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 5 | 1 | 1 | 1 | 1 | 3 | 3
hours | 2.00 [2.00 to 2.00] | 1.00 [1.00 to 1.00] | 10.00 [10.00 to 10.00] | 1.13 [1.13 to 1.13] | 1.82 [1.08 to 3.97] | 3.70 [2.00 to 9.70] | 1.92 [1.92 to 1.92] | 3.17 [3.17 to 3.17] | 4.00 [4.00 to 4.00] | 4.05 [4.05 to 4.05] | 3.00 [1.07 to 6.20] | 3.15 [2.07 to 3.87]

3. Secondary Outcome: Half-life Time From Overall Study
Description: as for outcome 2
Time Frame: 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 1&28
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Half-life Time Day 1:50mg; Half-life Time Day 1: 100 mg; Half-life Time Day 1: 200mg; Half-life Time Day 1: 300mg; Half-life Time Day 1: 450 mg; Half-life Time Day 1: 600 mg; Half-life Time Day 28: 50mg; Half-life Time Day 28:100 mg; Half-life Time Day 28: 200 mg; Half-life Time Day 28: 300 mg; Half-life Time Day 28: 450 mg; Half-life Time Day 28: 600mg: The time of plasma concentration drops from maximum to half
Arm/Group | Half-life Time Day 1:50mg | Half-life Time Day 1: 100 mg | Half-life Time Day 1: 200mg | Half-life Time Day 1: 300mg | Half-life Time Day 1: 450 mg | Half-life Time Day 1: 600 mg | Half-life Time Day 28: 50mg | Half-life Time Day 28:100 mg | Half-life Time Day 28: 200 mg | Half-life Time Day 28: 300 mg | Half-life Time Day 28: 450 mg | Half-life Time Day 28: 600mg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 5 | 1 | 1 | 1 | 1 | 3 | 3
hours | 2.42 | 1.30 | 4.33 | 1.93 | 2.38 (1.34) | 3.07 (1.52) | 1.60 | 2.34 | 1.41 | 2.11 | 1.81 (0.66) | 2.55 (1.30)

4. Secondary Outcome: Maximum Plasma Concentration After on Day 1
Description: Pharmacokinetic samples will be obtained from all the patients in each dose cohort treated in all phases of the study. Patients will only be sampled during their first treatment cycle only.
Time Frame: 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 1
Population: Pharmacokinetic (PK) Population: All patients who received at least 1 dose of antroquinonol with sufficient post-dose bio-samples collected for PK profile characterization.
Measure: Mean (95% Confidence Interval); unit: Log(mg/ml)
Groups:
- Cmax Day 1: the observed maximum plasma concentration after dosing on Day 1
Arm/Group | Cmax Day 1
Number analyzed (Participants) | 13
Log(mg/ml) | 0.504 [0.17 to 0.83]

5. Secondary Outcome: Maximum Plasma Concentration After Dosing on Day 28
Description: as for outcome 4
Time Frame: 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 28
Measure: Mean (95% Confidence Interval); unit: log(mg/ml)
Groups:
- Cmax Day 28: the observed maximum plasma concentration after dosing on Day 28
Arm/Group | Cmax Day 28
Number analyzed (Participants) | 10
log(mg/ml) | 0.682 [0.08 to 1.28]

6. Secondary Outcome: AUC0-t on Day 1
Description: as for outcome 4
Time Frame: within 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 1
Measure: Mean (95% Confidence Interval); unit: log(mg*hr/mL)
Groups:
- AUC0-t on Day 1: truncated area under the plasma concentration-time curve from the beginning of dosing to the last measurable concentration on Day 1
Arm/Group | AUC0-t on Day 1
Number analyzed (Participants) | 13
log(mg*hr/mL) | 0.641 [0.16 to 1.12]

7. Secondary Outcome: AUC0-t on Day 28
Description: as for outcome 4
Time Frame: 30 minutes prior to and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 14, and 24 hours after dose of Day 28
Measure: Mean (95% Confidence Interval); unit: log(mg*hr/mL)
Groups:
- AUC0-t on Day 28: truncated area under the plasma concentration-time curve from the beginning of dosing to the last measurable concentration on Day 28
Arm/Group | AUC0-t on Day 28
Number analyzed (Participants) | 10
log(mg*hr/mL) | 0.957 [0.59 to 1.32]

8. Secondary Outcome: Number of Participants in the PP Population With Better Than SD at Target Lesion, Better Than Non-CR/Non-PD at Non-target Lesion and no New Lesion
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for overall response by CT: Judgement by total siutation of target, non-target and new lesions.
  Meaning of Target lesion: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), Sum down 30% or more from target lesion baseline; Progressive Disease(PD), Sum up at least 20% from smallest value (nadir) and Absolute increase ≥ 5 mm; Stable Disease (SD), Neither enough shrinkage for PR nor enough growth for PD.
  non-target lesion: CR: All non-target lesions disappeared and All lymph nodes <10 mm; Non-CR/Non-PD: Non-target lesion(s) still present and Lymph nodes ≥10 mm; PD: Unequivocal progression; New lesion :Unequivocal new cancer lesions Overall SD response should be better than SD at target lesion, better than Non-CR/Non-PD t non-target lesion and no new lesion.
Time Frame: pre-screening and end of treatment
Population: Per-protocol (PP) Population: All patients who completed at least 3 cycles of treatment with proper imaging assessment (RECIST).
Measure: Number; unit: participants
Groups:
- Tumer Responce at Per-protocol (PP) Population: All patients who completed at least 3 cycles of treatment with proper imaging assessment (RECIST) of tumor size.
Arm/Group | Tumer Responce at Per-protocol (PP) Population
Number analyzed (Participants) | 3
participants | 3

9. Secondary Outcome: Safety Blood and Urine Test
Description: 1. Hematology laboratory data
  2. Biochemistry laboratory data
  3. Urinalysis
  4. AE; AE not including the natural progress of the underlying disease
  5. Incidence of toxicity ≥ grade 3 according to NCI CTCAE version 4.03
  6. Physical examination
  7. Vital signs changes
  8. Electrocardiogram examination results (including HR, QRS, QT, QTc, RR intervals)
Time Frame: pre-screenting and every 14-day period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: recorded immediatly as AE happen
Description: treatment-emergent adverse events (TEAEs) were reported as determined by the NCI CTCAE, Version 4.03. reported only related to the study drug
Arm/Group | Antroquinonol
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antroquinonol (N=13)
diarrhea (Gastrointestinal disorders) | 12 (12) — 12 patients, 92.3% [7 patients in grade 1, 53.8%, and 5 patients in grade 2, 38.5%]
vomiting (Gastrointestinal disorders) | 9 (9)
nausea (Gastrointestinal disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the PI should grand sponcer's agree to discuss or publish trial results after the trial is completed.